CLINICAL TRIAL: NCT02227277
Title: Towards Eradication: Reducing Proviral HIV DNA With Interferon-a Immunotherapy
Brief Title: Reducing Proviral HIV DNA With Interferon-a
Acronym: BEAT-HIV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Wistar Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Luis Montaner, Professor, Immunology Program and Director, HIV-1 Immunopathogenesis Laboratory, The Wistar Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES11990; 1U01AI110434 (NIH)
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: HIV; HIV/AIDS
Keywords: HIV; HIV-1; Pegintron; Peg-IFN-α2b; Viral suppression; ART cessation; Immune function; Innate immunity; Toxicity; Immune-based therapy; Treatment interruption; HIV Cure; HIV Eradication; BEAT-HIV; HIV Cure Trial; Cure Trial
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conditional 12-week ART interruption (Experimental): 18 participants will receive peg-IFN-α2b (1 μg/kg/week) for 20 weeks.
  Interventions: Drug: Peg-IFN-α2b
- Continuous ART (Experimental): 18 participants will receive peg-IFN-α2b (1 μg/kg/week) for 20 weeks.
  Interventions: Drug: Peg-IFN-α2b
- Control with continuous ART (No Intervention): 18 participants will continue their current ART regimens and be observed for 20 weeks.

INTERVENTIONS:
Drug: Peg-IFN-α2b — Arm 1: At week 4 of the treatment, ART will be interrupted. Viral load will be monitored every 2 weeks. ART will be resumed at the earlier of a) a single measurement of VL > 50 c/ml or b) 16 weeks of treatment, and subjects will be observed for the remaining 4 weeks (total of 20 weeks on treatment).
  Arm 2: In week 4, participants in arm 2 will add peg-IFN-α-2b to their ART regimen for a period of 20 weeks.
  Other Names: Pegintron
  Arms: Conditional 12-week ART interruption; Continuous ART

SUMMARY:
The purpose of this study is to determine if treatment with pegylated interferon alpha 2b (peg-IFN-α2b) will reduce the amount of integrated HIV DNA in peripheral blood cells and tissues of individuals with chronic HIV infection receiving antiretroviral treatment (ART).

A reduction and/or clearance of the latent viral reservoir (i.e.: virus that remains dormant in HIV-infected subjects receiving suppressive treatment ) is considered essential for HIV eradication.

By measuring the changes in integrated proviral HIV DNA, which is considered a surrogate measure of the latent reservoir, the investigators will establish if peg-IFN-α2b treatment should be considered as a component of future viral eradication strategies.

DETAILED DESCRIPTION:
Our long-term goal is to evaluate the effect of pegylated interferon (peg-IFN) α as an anti-HIV reservoir immunotherapy that could potentiate eradication strategies against HIV.

The present study is a 3-arm randomized clinical trial (RCT). The aim of this study is to determine whether a 20-week treatment course with 1μg/kg/week of pegylated interferon alpha 2 b (peg-IFN-α2b) will reduce the levels of HIV-1 proviral DNA levels in circulating PBMC and mucosa-associated lymphoid tissue (MALT) in HIV-infected individuals receiving long-term ART.

In addition, we will study if a 4-week interruption of ART is necessary to observe any change in proviral DNA levels.

In our previous study (NCT00594880) with a different form of Interferon alpha (peg-IFN-α2a), we observed a reduction in proviral DNA in peripheral blood cells in 50% of the patients. However, we did not measure the levels in MALT, and we could not determine whether or not an interruption of ART was necessary. The present study will address these questions.

We will also seek to determine the biological mechanisms (such as an increase in Natural Killer cell cytotoxicity) that mediate the antiviral effects of peg-IFN-α.

ELIGIBILITY:
Inclusion criteria

* 18-65 years of age
* Body weight ≥ 125 and ≤ 300 lbs
* Confirmed diagnosis of HIV-1 infection by western blot or by a documented HIV-1 viral load at screening.
* Currently receiving ART and on ART for ≥ 1 year
* VL < 50 copies/ml for ≥ 1 year, with at least 2 measurements in the previous year. 1 viral "blip" with VL< 400 copies/ml allowed if 1 or more measurements of < 50 copies/ml are available no more than 3 months before and 3 months after the "blip" without change in ART
* HIV viral load of <50 copies/ml at screening.
* CD4 >450 cells/µL at screening.
* a negative electrocardiogram (EKG, see section 7.4) for: a) men >45 years or women > 55 years of age b) younger subjects of either sex with two risk factors for coronary artery disease [smoking, hypertension (BP >140/90 or on antihypertensive medications), low HDL (<40 mg/dl), family history of premature CHD (<55 yrs males/<65 females, c) subjects with a Framingham score > 15% (men) or 10% (women)

Exclusion criteria Current or prior medications

* Confirmed clinical history of developing resistance to ART regimens that resulted in treatment changes
* Receiving didanosine as part of the participant's ART regimen at the time of screening
* Ongoing treatment with Isoniazid, Pyrazinamide, Rifabutin, Rifampicin, Ganciclovir, Valgancyclovir, Oxymetholone, Thalidomide or Theophylline.
* Ongoing treatment with anticoagulants
* Use of any investigational drug within 30 days prior to screening
* History or current use of immunomodulatory therapy for over 2 weeks during the 6 months prior to enrollment, including, but not limited to: IFN-α or γ (recombinant or pegylated), systemic corticosteroids (inhaled steroids allowed at the discretion of the Investigator); systemic cancer chemotherapy/irradiation; cyclosporin; tacrolimus (FK-506); OKT-3; any Interleukin, including IL-2; cyclophosphamide; methotrexate; IVIG (gamma globulin); G/M-CSF; hydroxyurea; thalidomide; pentoxifylline; thymopentin; thymosin; dithiocarbonate; polyribonucloside.
* History of adverse or allergic reactions to any type-1 interferon (e.g. IFN-α2a, IFN-α2b, IFN-β)

Current or prior clinical conditions

* History of severe depression, including history of suicidal ideation or attempt, or ongoing moderate depression determined by PHQ-9 at screening
* Type I diabetes mellitus, or type II diabetes mellitus that is not controlled with oral agents and/or insulin (i.e.: subjects with a history of diabetes mellitus and HA1C of > 9 in the last 3 months or at screening).
* Prior diagnosis of multiple sclerosis or other neurodegenerative disorders
* Significant co-existing lab abnormalities including: a) Anemia (Hgb <9.1 mg/dl men, <8.9 mg/dl women); b) Ongoing coagulopathy/clotting disorder; c) WBC <2000 cells/µl; d) Absolute neutrophil count (ANC) <1200 cells/ µl; e) Platelet count <60,000 cells/ µl; f) Liver disease (AST/ALT > 2.5x OR total bilirubin > 1.5x upper limits of norm (ULN), (if not receiving atazanavir) or direct bilirubin > 0.6 (if receiving atazanavir); g) Pancreatic disease (amylase : > 1.5 ULN, lipase > 1.5 ULN, triglycerides > 750 mg/dl); h Renal disease (creatinine > 2x ULN or creatinine clearance <60mg/dl (by Crockoff-Gault)
* Chronic HCV infection (HCV viremia), or HBV Ag positive and/ or HBV viremia (Notice: subjects with prior HCV infection with a documented sustained virologic response with treatment finishing >1 year prior to screening are eligible for enrollment).
* Liver cirrhosis or hepatic decompensation with Child Pugh score > 6
* History of major organ transplantation with an existing functional graft.
* Evidence of OI or other active infectious diseases or active malignancies
* Active Autoimmune diseases, including autoimmune hepatitis
* History of retinopathy or clinically significant ophthalmologic disease on eye exam performed within 60 days prior to initiation of IFN
* Significant EKG abnormalities (see section 7.4)

Other conditions

* Pregnancy or breastfeeding
* A planned pregnancy during study participation
* Lack of one of three strategies for birth control during study participation: a) Barrier contraceptives (male or female condoms with or without a spermicidal agent, diaphragm or cervical cap with spermicidal); b) Non-hormonal Intrauterine Devices (IUDs); c) Hormonal-based, including hormonal IUDs, in combination with barrier contraceptives.
* Body weight < 125 lbs or > 300 lbs
* Other conditions, such as active drug/alcohol abuse or dependence,that in the opinion of the Investigator would interfere with study compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-07-24 (Estimated)

PRIMARY OUTCOMES:
Integrated HIV proviral DNA | 24 weeks
  The study endpoint is the change in the number of copies of integrated HIV DNA/10^6 CD4+ T cells (as assessed by Alu-HIV gag PCR) between baseline and 20 weeks of peg-IFNα-2b administration (study week 24).

SECONDARY OUTCOMES:
Integrated proviral DNA in tissue | 24 weeks
  Copies of HIV DNA per tissue derived 2x106 isolated lymphocytes (GALT biopsy)-recovered lymphocyte (week 0 vs. week 24)
CD4 count | 24 weeks
  compare the frequency of occurrence of CD4 count < 350 (trigger to resume ART during ART interruption in arm 1) between study arms
Viral load | 24 weeks
  compare the frequency of occurrence of VL > 50 copies/ml (trigger for resuming ART during ART interruption in arm 1) between arms

OTHER OUTCOMES:
SUSAR (serious unexpected suspected adverse reactions) | 24 weeks
  compare occurrence of SUSAR between arms

CONTACTS AND LOCATIONS:
Overall Officials: Luis J. Montaner, DVM, DPhil, Principal Investigator — The Wistar Institute
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn-Presbyterian Hospital, Philadelphia, Pennsylvania
  - Jonathan Lax Center at Philadelphia FIGHT, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Azzoni L, Foulkes AS, Papasavvas E, Mexas AM, Lynn KM, Mounzer K, Tebas P, Jacobson JM, Frank I, Busch MP, Deeks SG, Carrington M, O'Doherty U, Kostman J, Montaner LJ. Pegylated Interferon alfa-2a monotherapy results in suppression of HIV type 1 replication and decreased cell-associated HIV DNA integration. J Infect Dis. 2013 Jan 15;207(2):213-22. doi: 10.1093/infdis/jis663. Epub 2012 Oct 26. PMID 23105144
- [Background] Mexas AM, Graf EH, Pace MJ, Yu JJ, Papasavvas E, Azzoni L, Busch MP, Di Mascio M, Foulkes AS, Migueles SA, Montaner LJ, O'Doherty U. Concurrent measures of total and integrated HIV DNA monitor reservoirs and ongoing replication in eradication trials. AIDS. 2012 Nov 28;26(18):2295-306. doi: 10.1097/QAD.0b013e32835a5c2f. PMID 23014521
- [Background] Sun H, Buzon MJ, Shaw A, Berg RK, Yu XG, Ferrando-Martinez S, Leal M, Ruiz-Mateos E, Lichterfeld M. Hepatitis C therapy with interferon-alpha and ribavirin reduces CD4 T-cell-associated HIV-1 DNA in HIV-1/hepatitis C virus-coinfected patients. J Infect Dis. 2014 May 1;209(9):1315-20. doi: 10.1093/infdis/jit628. Epub 2013 Nov 25. PMID 24277743
- [Derived] Papasavvas E, Azzoni L, Kossenkov AV, Dawany N, Morales KH, Fair M, Ross BN, Lynn K, Mackiewicz A, Mounzer K, Tebas P, Jacobson JM, Kostman JR, Showe L, Montaner LJ. NK Response Correlates with HIV Decrease in Pegylated IFN-alpha2a-Treated Antiretroviral Therapy-Suppressed Subjects. J Immunol. 2019 Aug 1;203(3):705-717. doi: 10.4049/jimmunol.1801511. Epub 2019 Jun 28. PMID 31253727
- See also: Montaner Lab at the Wistar Institute — http://www.wistar.org/our-science/scientists/luis-montaner-dvm-dphil
- See also: Infectious Disease Services at Penn-Presby — http://www.pennmedicine.org/infectious/presby/
- See also: Philadelphia FIGHT — https://fight.org